CLINICAL TRIAL: NCT02119546
Title: Effects of Exercise Training in Patients With Mild Cognitive Impairment and Early Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 200912126R
Record Dates: First submitted 2012-11-19; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Mild CognitIve Impairment; Alzheimer's Disease
Keywords: Mild CognitIve impairment; Alzheimer's disease; Cognitive function; Exercise training
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Exercise; Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise intervention (Experimental): Aerobic exercise and dual-task training
  Interventions: Other: Aerobic exercise
- Stretch exercise (Active Comparator): Stretch exercise & sitting balance
  Interventions: Other: Stretch exercise

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise and dual-task training
  Arms: Exercise intervention
Other: Stretch exercise — Stretch exercise & sitting balance
  Arms: Stretch exercise

SUMMARY:
The purposes of this study are:

1. To investigate whether a 3-month exercise training program would improve cognitive function, motor performance, integrity of brain fiber tracts and cerebral blood flow;
2. To investigate the possible neuro-anatomical and neurophysiological mechanisms of exercise training on cognitive function, motor performance, integrity of brain fiber tract and cerebral blood flow in patients with mild cognitive impairment and in those with early Alzheimer's disease;
3. To investigate the influence of different apolipoprotein E (APOE) genotypes on the above-mentioned exercise effects.

The results of this study will provide medical evidence for the effects of exercise training on mild cognitive impairment and on early Alzheimer's disease; and will provide understanding of the mechanisms mediating these effects. More importantly, the results serve as the basis for future larger-scale exercise clinical trials for these two patient populations.

DETAILED DESCRIPTION:
Recent studies have shown that exercise training could decrease the risk of dementia in the elderly population. Exercise training could also slow down the speed of deterioration of memory and other cognitive functions in patients who already have mild cognitive impairment or early Alzheimer's disease. However, the mechanisms of such effects are still unknown. Whether exercise training could improve neural fiber integrity, blood flow, or motor performance of these patients also remain unexplored.

Therefore, the purposes of this study are:

1. To investigate whether a 3-month exercise training program would improve cognitive function, motor performance, integrity of brain fiber tracts and cerebral blood flow;
2. To investigate the possible neuro-anatomical and neurophysiological mechanisms of exercise training on cognitive function, motor performance, integrity of brain fiber tract and cerebral blood flow in patients with mild cognitive impairment and in those with early Alzheimer's disease;
3. To investigate the influence of different APOE genotypes on the above-mentioned exercise effects.

We will conduct a single-blinded, randomized controlled clinical trial. We will recruit 60 patients with mild cognitive impairment or early Alzheimer's disease. The participants will be randomly classified into the exercise training group or control group. The exercise training group will receive health education and exercise training of moderate intensity, 3 times a week, for 12 weeks. The control group will receive health education only. Both groups will receive pre- (week 0), post- (week 12), and follow-up (week 24 after the end of the program) examinations for cognitive function, motor performance, diffusion tensor or diffusion spectrum magnetic resonance imaging, and transcranial duplex. We will compare the group differences on the aforementioned outcome measures brought by 12-week exercise training. We will also perform analysis of the correlations between the changes in these outcome measures to explore the possible neural or physiological mechanisms mediating the training effects. The effects of different APOE genotypes on these outcome measures will also be compared.

The results of this study will provide medical evidence for the effects of exercise training on mild cognitive impairment and on early Alzheimer's disease; and will provide understanding of the mechanisms mediating these effects. More importantly, the results serve as the basis for future larger-scale exercise clinical trials for these two patient populations.

ELIGIBILITY:
Inclusion Criteria:

* 45~85 years old and had independent walking ability
* The MCI is diagnosed basically on Petersen's criteria (Petersen, 2001), CDR score of 0.5 but normal activity of daily living /instrumental activities of daily living, and not demented
* Diagnosis of Alzheimer's disease based on NINCDS-ADRDA criteria for probable Alzheimer disease (McKhann, et al., 1984)

Exclusion Criteria:

* The subjects who had any neurological, musculoskeletal, cardio-pulmonary disorder which would cause gait disorder or cognitive dysfunction such as stroke, Parkinson disease, or arthritis were excluded

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-05; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Color Trails Test at week12 and Week24 | Baseline, Week12, Week24
  To investigate the cognitive executive function

SECONDARY OUTCOMES:
Change from baseline in walking speed at week12 and Week24 | baseline, week12 and Week24
  To investigate walking ability

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Jang Chiu, PhD, Study Chair — Neurology department, National Taiwan University Hospital; Yu-Hsiu Chu, PhD, Principal Investigator — Department of Physical Therapy, China Medical University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan